CLINICAL TRIAL: NCT07099443
Title: Determinants of the Response to BTK Degraders (BTKd) in Double Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: Determinants of the Response to BTK Degraders (BTKd) in Double Refractory CLL
Acronym: REBELLE
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC25_0135
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Bruton tyrosine kinase inhibitors; BCL-2 inhibitors; BTK degraders
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples, additional bone marrow samples, and leftover lymph node tissue obtained during procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- double-refractory CLL patients: Collection of additional samples of blood and bone marrow or residual lymph node biopsy at the time of inclusion (for diagnosis or relapse) and relapse.
  Interventions: Other: Non-Interventional Sample Collection and Analysis

INTERVENTIONS:
Other: Non-Interventional Sample Collection and Analysis — This study is observational. Biological samples are collected as part of standard care or for research purposes and analyzed to characterize resistance mechanisms. No treatment or intervention is administered as part of the study protocol.

SUMMARY:
The aim of the REBELLE cohort - bio-collection is to collect samples from patients with Chronic Lymphocytic Leukemia (CLL), to facilitate access for the National Institute of Health and Medical Research (INSERM) to patients with double-refractory CLL. To do this, an additional blood or bone marrow sample to those planned in the context of patient care or a residual lymph node biopsy sample will be collected after signing consent. These samples will first be sent to the Filothèque for temporary storage, and will then be transferred to CRCI²NA (Nantes - Angers Cancer and Immunology Research Center) for analysis with the aim of studying the mechanisms of resistance and response to BTK degraders (BTKd).

DETAILED DESCRIPTION:
Chronic Lymphocytic Leukemia (CLL) is a malignant B-cell disorder characterized by the accumulation of CD19+CD5+ lymphocytes in the bone marrow, lymph nodes, spleen, and peripheral blood. It has an incidence of approximately 4.2 cases per 100,000 people annually, with a median diagnosis age of 72 years. CLL exhibits marked biological and clinical heterogeneity, influenced by prognostic factors such as Immunoglobulin Heavy Chain Variable Region (IGHV) mutation status, TP53 alterations, and complex karyotypes. The disease is typically indolent, and treatment initiation follows criteria established by the International Workshop on CLL (IWCLL). Symptoms, when present, include lymphadenopathy, cytopenias, and infections. About one-third of patients require treatment at diagnosis, another third within ten years, and the remaining third may never need therapy. Although incurable, CLL generally has favorable progression-free and overall survival rates.Historically, chemotherapy was the main treatment, but the advent of targeted oral therapies-particularly Bruton tyrosine kinase inhibitors (BTKi) and BCL-2 inhibitors (BCL-2i)-has significantly improved patient outcomes. BTKi block the BTK enzyme critical for B-cell receptor signaling, thereby inhibiting malignant B-cell proliferation and survival. BCL-2 inhibitors induce apoptosis by binding to the anti-apoptotic BCL-2 protein, which CLL cells often overexpress. Combined use of these agents with monoclonal antibodies has become standard care. Despite these advances, approximately 20% of patients develop resistance to chemotherapy or targeted therapies. A rare but clinically significant subgroup, termed double refractory, fails to respond to both BTKi and BCL-2i and has a poor prognosis. Defining resistance includes clinical progression on therapy and biological markers such as mutations associated with drug resistance. Resistance to BTKi arises from compensatory signaling pathways or mutations within BTK, whereas resistance to BCL-2 inhibitors is typically identified when patients relapse during or soon after treatment.. To overcome resistance to BTKi, novel BTK degraders (BTKd) are under development. Unlike BTKi, these heterobifunctional molecules induce proteasomal degradation of the BTK protein via ubiquitination, showing promising preclinical efficacy. However, limited clinical data exist on BTKd, and researchers still need to carry out a full evaluation of their effectiveness against other resistance mechanisms and in combination with current immunotherapies. To gain a better understanding of resistance and response to BTKd, establishing a dedicated cohort and biobank of samples from double-refractory CLL patients is essential. Collaborating with research teams specialized in hematologic malignancies, such as the CRCI²NA group, and leveraging existing frameworks like the FILO/LYSA ( French Innovative Leukemia Organization/Network for clinical lymphomas and CLL/WM research) networks, will enable comprehensive translational studies. This initiative aims to address the urgent need for novel therapeutic strategies in this challenging patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed double refractory CLL to both BTKi and BCL-2i, defined as:

  * Any patient who has received both a BTKi and a BCL-2i, regardless of treatment regimen, and has shown clinical progression either during treatment with both BTKi and BCL-2i, or within 36 months after stopping BCL-2i.
  * Any patient identified with known biological resistance mutations to BTKi or BCL-2i, regardless of clinical progression.
* Patient who has provided informed consent to participate in the study.
* Patient covered by a social security health insurance plan

Exclusion Criteria:

* Minor patients.
* Adults under guardianship.
* Protected persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Double refractory CLL patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2039-09-15 (Estimated); Study Completion 2039-09-15 (Estimated)

PRIMARY OUTCOMES:
Characterization of resistance mechanisms to BTK degraders in double-refractory CLL patients | Up to 5 years after inclusion
  The primary outcome is the in-depth characterization of tumor cells and their microenvironment in double-refractory CLL patients. Analyses will be performed using cellular biology (e.g., flow cytometry), molecular biology (e.g., RNA sequencing), and bioinformatics (e.g., deconvolution). Functional studies include the development of preclinical ex vivo models (2D/3D culture) and gene editing of primary cells using CRISPR/Cas9 technology, based on the expertise of Team 11 at CRCI²NA.
  The study will include 60 patients over a 9-year enrollment period. Each participant will be followed for 5 years, resulting in a total study duration of 14 years.

SECONDARY OUTCOMES:
Development of preclinical ex vivo culture models | Up to 5 years after inclusion
  Establishment of 2D and 3D ex vivo culture systems using primary CLL cells to replicate tumor behavior and evaluate functional characteristics.
Genetic modification of primary CLL cells | Up to 5 years after inclusion
  Application of gene editing technologies (e.g., CRISPR/Cas9) to modify primary chronic lymphocytic leukemia cells in order to investigate gene function and resistance pathways.
Genomic data analysis to identify resistance-related genes | Up to 5 years after inclusion
  Comprehensive genomic and transcriptomic profiling of CLL samples to identify genetic alterations and expression patterns associated with resistance to BTK degraders.
Identification of new tumor targets | Up to 5 years after inclusion
  Discovery and validation of novel molecular targets involved in tumor survival and drug resistance in CLL using omics data and functional assays.
Pharmacological targeting of novel candidate molecules | Up to 5 years after inclusion
  Functional validation of newly identified targets through pharmacological inhibition to assess their therapeutic potential in vitro using CLL models.
Generation of knockout cell lines for genes of interest | Up to 5 years after inclusion
  Creation of gene knockout models in CLL cell lines via CRISPR/Cas9 to explore the biological role of specific resistance-associated genes.
Generation of drug-resistant cell lines and comparative RNA sequencing | Up to 5 years after inclusion
  Development of CLL cell lines resistant to BTK degraders followed by RNA sequencing analysis to compare gene expression profiles with drug-sensitive lines.
Reconstruction of the tumor microenvironment using co-culture systems | Up to 5 years after inclusion
  Establishment of co-culture models including immune (T lymphocytes, nurse-like cells) and/or stromal cells (from lymph nodes or bone marrow) to mimic the CLL tumor microenvironment.

CONTACTS AND LOCATIONS:
Overall Officials: Anne LOK, MD, PhD, Principal Investigator — Hospital of Nantes
Locations (14):
- France (14):
  - CHU de Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Institut Bergonié, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHD Vendée, La Roche-sur-Yon
  - Centre Léon Bernard, Lyon
  - Institut Paoli-Calmettes (Marseille), Marseille
  - CHU de Montpellier, Montpellier
  - CH Régional Universitaire de Nancy, Nancy
  - University Hospital, Nantes
  - Hôpital Avicenne (AP-HP), Paris
  - Hôpital Universitaire Pitié Salpêtrière de Paris, Paris
  - CHU de Poitiers, Poitiers
  - Centre Henri-Becquerel de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: Undecided